CLINICAL TRIAL: NCT05173025
Title: Effect of Fimasartan or Amlodipine on Extended Renin-angiotensin System in Patients With Type 2 Diabetes and Hypertension
Brief Title: Effect of Fimasartan on Extended RAS and Vascular Functions in Patients With Type 2 Diabetes and Hypertension
Acronym: FAoRAS
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Seoul National University Bundang Hospital (Other)
Responsible Party: Principal Investigator, Soo Lim, Professor, Seoul National University Bundang Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: B-1606-351-003
Record Dates: First submitted 2021-12-27; First posted 2021-12-29 (Actual); Last update posted 2023-08-14 (Actual); Status verified 2023-08

CONDITIONS: Hypertension; Atherosclerosis; Diabetes Mellitus, Type 2; Renin Hypertension
MeSH Terms: conditions — Hypertension; Atherosclerosis; Diabetes Mellitus, Type 2 | interventions — fimasartan

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fimasartan (Experimental): - Fimasartan group: Fimasartan, 60 mg once a day, oral administration
  Interventions: Drug: Fimasartan
- Amlodipine (Active Comparator): - Comparator group: Amlodipine, 5 mg once a day, oral administration
  Interventions: Drug: Fimasartan

INTERVENTIONS:
Drug: Fimasartan — - Fimasartan group: fimasartan, 60 mg once a day, oral administration
  Other Names: Kanarb

SUMMARY:
In this study, we will assess the change of extended renin-angiotensin system including serum ACE-2 and angiotensin(1-7) levels and subclinical atherosclerosis after using fimasartan (an ARB), compared to amlodipine in hypertensive patients with T2DM.

DETAILED DESCRIPTION:
Several clinical trials aimed at studying the benefits of RAS blockade in the diabetic complications. HOPE, RENAAL, IRMA2, IDNT, ONTARGET studies proved that ACE inhibitors or ARBs reduced the risk of diabetic complications.

Recent studies proved that fimasartan, one of the ARBs, stabilizes the activity of renin-angiotensin system. However, understanding the change in concentration of serum ACE, ACE-2, angiotensin(1-7), and angiotensin-II should help clinicians select more appropriate drug between ACE inhibitors and ARBs with clear evidence. Moreover, since RAS antagonists are the first-line drugs for antihypertensive therapy in patients with T2DM, it is meaningful to understand the change of RAS-related factors in serum after using the drugs.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 30 years old
* Type 2 diabetes by American Diabetes Association criteria
* HbA1c: 6.5% ≤ - < 10.0%
* Systolic blood pressure: 140 ≤ - < 180 mmHg or Diastolic blood pressure: 85 ≤ - < 110 mmHg
* Statin (-) or no change in low to moderate intensity statin [14] dose in recent 3 months

Exclusion Criteria:

* Contraindication of fimasartan or amlodipine
* History of RAS inhibitors (ACE inhibitors or ARBs) or calcium channel blockers in the previous 3 months
* Pregnant women, women with potential of pregnancy not using adequate contraception method as evaluated by the investigator, lactating women
* Type 1 diabetes or diabetes secondary to chronic pancreatitis or to pancreatectomy
* Confirmed cardiovascular disease (acute coronary syndrome, stroke, or transient ischemic attack) within 3 months of screening
* Chronic hepatitis B or C (except healthy carrier of HBV), liver disease (AST/ALT > 3-fold the upper limit of normal)
* Chronic kidney disease (serum creatinine > 2.0 mg/dL)
* Hyperkalemia serum potassium >5.0 mEq/L
* Any previous cancer within 5 years (except squamous cell cancer, cervical cancer, thyroid cancer with appropriate treatment) except thyroid cancer or carcinoma in situ

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2018-01-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Angiotensin(1-7) | 12 weeks
  Changes of serum angiotensin(1-7) at week 12 from baseline

SECONDARY OUTCOMES:
Blood pressure | 12 weeks
  Change in blood pressure from baseline to week 12
  Change in blood pressure from baseline to week 24
  Change in blood pressure from baseline to week 24
ACE-2 | 12 weeks
  Change in ACE-2 from baseline to week 12
  Change in blood pressure from baseline to week 24
  Change in blood pressure from baseline to week 24
ACE | 12 weeks
  Change in ACE from baseline to week 12
  Change in blood pressure from baseline to week 24
  Change in blood pressure from baseline to week 24
Renin | 12 weeks
  Change in renin from baseline to week 12
  Change in blood pressure from baseline to week 24
  Change in blood pressure from baseline to week 24
angiotensin | 12 weeks
  Change in angiotensin from baseline to week 12
  Change in blood pressure from baseline to week 24
  Change in blood pressure from baseline to week 24
atherosclerosis | 12 weeks
  Change in atherosclerosis from baseline to week 12
  Change in blood pressure from baseline to week 24
  Change in blood pressure from baseline to week 24
Muscle mass | 12 weeks
  Change in muscle mass from baseline to week 12
  Change in blood pressure from baseline to week 24
  Change in blood pressure from baseline to week 24
Fat mass | 12 weeks
  Change in fat mass from baseline to week 12
  Change in blood pressure from baseline to week 24
  Change in blood pressure from baseline to week 24
HbA1c | 12 weeks
  Change in HbA1c from baseline to week 12
  Change in blood pressure from baseline to week 24
  Change in blood pressure from baseline to week 24

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: No